CLINICAL TRIAL: NCT04900805
Title: Studies of Physiological Effects During Practices of Alternative Mediicine
Brief Title: Temperature Variation During Meditative Practices
Status: Completed | Type: Observational
Sponsor: Istituto Nazionale Biostrutture e Biosistemi (Other)
Responsible Party: Sponsor
Other Study IDs: INBB1705
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The temperature on selected points of the hands has been monitored during meditative practices. The practitioner is in complete rest for the time of the measure, and only mental activity is carried out. The purpose is to verify if the heat sensation, that is normally felt, is a real, measurable physiological effect, or if it is just a subjective feeling. Quantitative data analysis is foreseen.

DETAILED DESCRIPTION:
Qigong is a traditional Chinese method for wellness and healing. During practice, which is based on the Qi circulation, it is usual to feel warmth, especially at the hands. The main purpose of this study is to verify if the sensation of heat is not just a subjective feeling but is a real, measurable physiological effect. Quantitative information will be hopefully derived from a simple data analysis. The study will be extended also to deep prayer meditation.

The measurement sessions will consist of two periods of practice separated by one pause period, to ensure that the temperature variation is not due to spurious effects.

T type thermocouples will be used for the temperature measurements, with sensors in the form of small copper disk. The thermocouples will be connected to a data logger, and the results analyzed. The sensors will be positioned in different points of the hands, either on the palm and on the dorsum. The Laogong (PC8) acupuncture point will be preferentially chosen, because is a very important point, from the energetic point of view, of the Traditional Chinese Medicine. and because the sensation of heat is more acute in this point. Other points will be also measured, and compared with the Laogong.

ELIGIBILITY:
Inclusion Criteria:

. Experience in meditative practice

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with experience in meditative practice
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-19 (Actual)

PRIMARY OUTCOMES:
Temperature variation during meditative practice | 1 hour
  The variation of the temperature in specific points of the hands will be obtained during meditative practice. In general the study will consist in two periods of practice separated by a pause

SECONDARY OUTCOMES:
Comparison of temperature variation in different points of the hands | 1 hour
  The temperature will be measured in different points of the hands, in relation with relevant points of the Traditional Chines medicine (Acupuncture points), and their behavior compared

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Lagomarsino, Principal Investigator — Istituto Nazionale Biostrutture e Biosistemi
Locations (1):
- INBB, Roma, Italy